CLINICAL TRIAL: NCT02851069
Title: Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C - An Observational Study in Colombia (outCome)
Brief Title: Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C in Colombia
Acronym: outCome
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-024
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-05

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Paritaprevir/r - Ombitasvir, ± Dasabuvir; Sustained Virological Response; Observational Study; Chronic Hepatitis C genotype 1
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Hepatitis C Virus Genotype 1 (HCV + GT1): ABBVIE REGIMEN (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg once daily] with or without dasabuvir [250 mg twice daily]), and with or without weight-based ribavirin (± RBV; dosed 1,000 or 1,200 mg daily divided twice a day) for 12 or 24 weeks in HCV + GT1 participants.

SUMMARY:
This is a prospective, multi-center observational study in adult participants chronically infected with hepatitis C virus (HCV) receiving the interferon-free ABBVIE REGIMEN (ombitasvir/paritaprevir/ritonavir with or without dasabuvir) with or without ribavirin (RBV). The prescription of a treatment regimen was at the discretion of the physician in accordance with local clinical practice and label.

This study focused on collecting real world data. Follow-up visits, treatment, procedures and diagnostic methods followed physicians' routine clinical practice using a 12-week treatment regimen (four visits plus two interim data collection windows) or a 24-week treatment regimen (four visits plus three interim data collection windows) and is based on the anticipated regular follow-up for patients undergoing treatment for chronic hepatitis C (CHC). Participants are observed for the duration of the ABBVIE REGIMEN therapy and for up to 24 weeks after treatment completion.

DETAILED DESCRIPTION:
This prospective, multi-center observational study in adult participants chronically infected with hepatitis C virus (HCV), receiving the interferon-free ABBVIE REGIMEN with or without RBV are offered the opportunity to participate in this study during a routine clinical visit at the participating sites at the discretion of the physician and is made independently from this observational study and preceded the decision to offer the participant the opportunity to participate in this study.

After written informed consent is obtained, demographics, HCV disease characteristics, co-morbidities, co-medication, treatment details, and laboratory assessments as recorded in the participant's medical records (source documentation) are documented in the electronic case report form (eCRF). Participants are observed for the duration of the ABBVIE REGIMEN therapy and for up to 24 weeks after treatment completion. No patient identifiable information was captured; a unique participant number was automatically allocated by the web based system once the investigator or designee created a new participant file.

This study focuses on collecting real world data. Follow-up visits, treatment, procedures and diagnostic methods follow physicians' routine clinical practice. The observational study period entailed the following data collection schemes:

* 12-week treatment regimen: four visits plus two interim data collection windows
* 24-week treatment regimen: four visits plus three interim data collection windows This schedule was based on the anticipated regular follow-up for patients undergoing treatment for CHC.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve or -experienced adult male or female participants with confirmed CHC, genotype 1, receiving combination therapy with the interferon-free ABBVIE REGIMEN (ombitasvir/paritaprevir/ritonavir with or without dasabuvir) ± ribavirin (RBV) according to standard of care and in line with the current local label.
* If RBV is co-administered with the ABBVIE REGIMEN , it has been prescribed in line with the current local label (with special attention to contraception requirements and contraindication during pregnancy).
* Participant must not be participating or intending to participate in a concurrent interventional therapeutic trial.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic hepatitis C (CHC), genotype 1, receiving combination therapy with the interferon-free ABBVIE REGIMEN ± RBV.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (6):
- Colombia (6):
  - Fundacion Cardioinfantil, Bogotá
  - Cic Cali, Cali
  - Centro Medico lmbanaco de Cali I, Cali
  - Pharos Centro de Estudios Clin, Cartagena
  - IPS Medicos Internistas Del Ca I, Manizales
  - Fundacion Hospitalaria San Vin, Medellín

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ferenci P, Bourgeois S, Buggisch P, Norris S, Curescu M, Larrey D, Marra F, Kleine H, Dorr P, Charafeddine M, Crown E, Bondin M, Back D, Flisiak R. Real-world safety and effectiveness of ombitasvir/paritaprevir/ritonavir +/- dasabuvir +/- ribavirin in hepatitis C virus genotype 1- and 4-infected patients with diverse comorbidities and comedications: A pooled analysis of post-marketing observational studies from 13 countries. J Viral Hepat. 2019 Jun;26(6):685-696. doi: 10.1111/jvh.13080. Epub 2019 Mar 5. PMID 30739368

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 66 participants were enrolled in the study; 1 participant never started treatment and thus the safety population was comprised of 65 participants. In this study, the safety population, target population, and core population were identical.
Groups:
- ABBVIE REGIMEN ± Ribavirin (RBV): ABBVIE REGIMEN (ombitasvir/paritaprevir/ritonavir with or without dasabuvir), and with or without weight-based ribavirin (± RBV) for 12 or 24 weeks
Period: Overall Study
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Started (Received at least 1 dose of study drug.) | 65
Completed | 59
Not Completed | 6
Not completed — Failure to Return | 3
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: The Core Population (CP): defined as all participants of the target population (all participants in the safety population who met inclusion criteria) who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype).
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response at 12 Weeks (SVR12) Post-treatment
Description: SVR12 was defined as plasma hepatitis C virus (HCV) ribonucleic acid (RNA) level ˂50 IU/mL 12 weeks after end of treatment (EoT) (defined as after last actual dose of the ABBVIE REGIMEN [paritaprevir/ritonavir - ombitasvir ± dasabuvir] or ribavirin [RBV]).
Time Frame: 12 weeks (i.e. 70 to 126 days) after the last dose of study drug (up to 24 weeks)
Population: Core Population (CP): defined as all participants of the target population (all participants in the safety population who met inclusion criteria) who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 65
percentage of participants | 87.7 [77.5 to 93.6]

2. Secondary Outcome: Percentage of Participants With Virologic Response at End of Treatment (EoT)
Description: Virologic response is defined as HCV RNA level <50 IU/mL.
Time Frame: Up to EoT, maximum of 24 weeks
Population: CP
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 65
percentage of participants | 95.4 [87.3 to 98.4]

3. Secondary Outcome: Number of Participants Meeting Premature Study Drug Discontinuation
Description: Premature study drug discontinuation was defined as participants who prematurely discontinued study drug (ABBVIE REGIMEN or RBV) and who experienced no on-treatment virologic failure (defined as breakthrough [at least 1 documented HCV RNA ˂50 IU/mL followed by HCV RNA ≥50 IU/mL during treatment] or failure to suppress [each measured on-treatment HCV RNA value ≥50 IU/mL]).
Time Frame: Up to EoT, maximum of 24 weeks
Population: CP
Measure: Number; unit: participants
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 65
participants
  Premature Termination ABBVIE REGIMEN | 4
  No Premature Termination ABBVIE REGIMEN | 61

4. Secondary Outcome: Percentage of Participants Meeting Each and Any SVR12 Non-response Criteria
Description: For a participant to be include in this analysis, the participant needed to meet each and any of the following SVR12 non-response categories:
  * On-treatment virologic failure (breakthrough [defined as at least one documented HCV RNA <50 IU/mL followed by HCV RNA ≥50 IU/mL during treatment] or failure to suppress [each measured on-treatment HCV RNA value ≥50 IU/mL]);
  * Relapse (defined as HCV RNA <50 IU/mL at actual EoT followed by HCV RNA ≥50 IU/mL post-treatment for participants who completed treatment [not more than 7 days shortened]);
  * Premature study drug discontinuation with no on-treatment virologic failure;
  * Missing SVR12 data and/or none of the above criteria (including participants with missing SVR12 data).
  Abbreviations: EoT=end of treatment.
Time Frame: During treatment and 12 weeks (i.e. at least 70 days) after the last dose of study drug (up to 24 weeks)
Population: CP
Measure: Number; unit: percentage of participants
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 65
percentage of participants
  Non-response 12 weeks after EoT | 12.3
  On-treatment virologic failure | 1.5
  Relapse | 1.5
  Premature treatment discontinuation | 4.6
  Missing SVR12 data/None of the above criteria | 4.6

5. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse was defined as confirmed HCV RNA <50 IU/mL at EoT or at the last on-treatment HCV RNA measurement followed by HCV RNA ≥50 IU/mL post-treatment in participants who were treated.
Time Frame: 12 weeks (i.e. at least 70 days) after the last dose of study drug
Population: CP
Measure: Number; unit: percentage of participants
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 65
percentage of participants | 1.5

6. Secondary Outcome: Percentage of Participants With Relapse at EoT
Description: Relapse was defined as confirmed HCV RNA <50 IU/mL at EoT followed by HCV RNA ≥50 IU/mL post treatment in participants who completed treatment (actual duration of ABBVIE REGIMEN is not shortened more than 7 days) and had HCV RNA results available in the SVR12 window.
Time Frame: 12 weeks (i.e. at least 70 days) after the last dose of study drug
Population: CP of participants with EoT response whose last post-treatment HCV RNA test result did not show virologic response
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 57
percentage of participants | 1.8 [0.3 to 9.3]

7. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: Viral breakthrough was defined as at least 1 documented HCV RNA <50 IU/mL followed by HCV RNA ≥ 50 IU/mL during treatment.
Time Frame: Up to EoT, maximum of 24 weeks
Population: CP
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 65
percentage of participants | 0.0 [0.0 to 7.4]

8. Secondary Outcome: Percentage of Participants Meeting On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as breakthrough (at least 1 documented HCV RNA <50 IU/mL followed by HCV RNA≥ 50 IU/mL during treatment) or failure to suppress (each measured on-treatment HCV RNA value ≥50 IU/mL).
Time Frame: Up to EoT, maximum of 24 weeks
Population: CP
Measure: Number; unit: percentage of participants
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 65
percentage of participants | 1.5

9. Secondary Outcome: Percentage of Participants With Rapid Virologic Response at Week 4 (RVR4)
Description: RVR4 was defined as HCV RNA < 50 IU/mL at Week 4.
Time Frame: Week 4
Population: CP
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 65
percentage of participants | 66.2 [54.0 to 76.5]

10. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 24 Weeks (SVR24) After EoT
Description: SVR24 was defined as HCV RNA < 50 IU/mL 24 weeks after EoT. During the course of the study, standard of care was changing and it was no longer common practice to assess SVR24.
Time Frame: 24 weeks after EoT (up to 24 weeks)
Population: CP participants with an SVR24 assessment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 9
percentage of participants | 44.4 [18.9 to 73.3]

11. Other Pre Specified Outcome: EuroQol 5 Dimension 5 Level (EQ-5D-5L) Questionnaire Index Score: Change From Baseline to EoT
Description: The EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by participants. The 5 items in the questionnaire comprise 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on 5 levels of severity (1: indicating no problem, 2: indicating slight problems, 3: indicating moderate problems, 4: indicating severe problems, 5: indicating extreme problems), and a separate VAS. The higher the score, the worse the quality of life. For the VAS, the higher the score, the better the quality of life. Participant responses to the EQ-5D-5L were used to generate a health status index (HSI). HSI ranges is anchored at 0 (dead) and 1 (full health).
Time Frame: EoT (up to 24 weeks)
Population: CP participants contributing to summary statistics. Changes were only calculated for participants with non-missing assessments at both time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 53
units on a scale | 0.005 (0.143)

12. Other Pre Specified Outcome: EQ-5D-5L Questionnaire Index Score: Change From Baseline to 12 Weeks Post EoT
Description: The EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by participants. The 5 items in the questionnaire comprise 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) each of which are rated on 5 levels of severity (1: indicating no problem, 2: indicating slight problems, 3: indicating moderate problems, 4: indicating severe problems, 5: indicating extreme problems), and a separate VAS. The higher the score, the worse the quality of life. For the VAS, the higher the score, the better the quality of life. Participant responses to the EQ-5D-5L were used to generate a HSI. HSI ranges is anchored at 0 (dead) and 1 (full health).
Time Frame: 12 weeks post EoT (up to 24 weeks)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 54
units on a scale | 0.039 (0.122)

13. Other Pre Specified Outcome: EQ-5D-5L Questionnaire Index Score: Change From Baseline to 24 Weeks Post EoT
Description: as for outcome 12
Time Frame: 24 weeks post EoT (up to 24 weeks)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 22
units on a scale | 0.046 (0.111)

14. Other Pre Specified Outcome: EQ-5D-5L Questionnaire VAS: Change From Baseline to EoT
Description: The EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by participants. Participants also rated their perception of their overall health on a separate VAS. The scale is numbered from 0 to 100. The higher the score, the better the quality of life.
Time Frame: End of Treatment (up to 24 weeks)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 54
units on a scale | 5.7 (10.40)

15. Other Pre Specified Outcome: EQ-5D-5L Questionnaire VAS: Change From Baseline to 12 Weeks Post EoT
Description: as for outcome 14
Time Frame: 12 weeks post EoT (up to 24 weeks)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 53
units on a scale | 7.5 (16.12)

16. Other Pre Specified Outcome: EQ-5D-5L Questionnaire VAS: Change From Baseline to 24 Weeks Post EoT
Description: as for outcome 14
Time Frame: 24 weeks post EoT (up to 24 weeks)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 22
units on a scale | 4.0 (12.41)

17. Other Pre Specified Outcome: Number of Participants With Co-morbidities at Baseline (Day 0)
Description: Co-morbidities/co-infections were defined as hepatitis C virus (HCV) co-infections (human immunodeficiency virus [HIV] or hepatitis B virus [HBV], tuberculosis, schistosomiasis), liver/chronic hepatitis C (CHC) related co-morbidities (liver transplantation, hepatocellular carcinoma, non-alcoholic steatosis, alcoholic liver disease, primary biliary cirrhosis, auto-immune hepatitis, Wilson disease, cryoglobulinemia, porphyria cutanea tarda, auto-immune skin disease), and other co-morbidities (chronic kidney disease, psychiatric disorders, diabetes mellitus, insulin resistance, metabolic syndrome, lipid disorder, cardiovascular disease, immunologically mediated disease, hyper-/hypothyroidism, hemophilia, Thalassemia, sickle cell anemia, V. Willebrand disease, psychoactive substance dependency, kidney transplant, or other).
Time Frame: Baseline (Day 0)
Population: CP
Measure: Number; unit: participants
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 65
participants
  All co-morbidities and co-infections | 58
  HCV Co-infections | 2
  Liver and/or CHC related co-morbidities | 5
  Other Co-morbidities | 57
  Kidney Transplantation | 3
  Chronic Kidney Disease | 7
  Psychiatric Disorders | 3
  Diabetes Mellitus | 14
  Lipid Disorder | 4
  Hypothyroidism | 17
  Cardiovascular disease | 28
  Hemophilia | 2
  Other | 40

18. Other Pre Specified Outcome: Number of Participants With Concomitant Medications
Description: This includes all participants that took at least 1 concomitant medication from the time when the decision was made to initiate treatment with the ABBVIE REGIMEN until after the last dose.
  Abbreviations: ACE= angiotensin-converting-enzyme; GERD=gastroesophageal reflux.
Time Frame: Day 0 to EoT, maximum 24 weeks
Population: Safety Population: defined as all enrolled participants who received at least one dose of the ABBVIE REGIMEN
Measure: Number; unit: participants
Arm/Group | ABBVIE REGIMEN ± Ribavirin (RBV)
Number analyzed (Participants) | 65
participants
  Number taking at least 1 co-medication | 55
  Beta Blocking Agents | 18
  Thyroid Therapy | 17
  Vitamins | 16
  Angiotensin II Antagonists | 15
  Drugs for Peptic Ulcer and GERD | 13
  Blood glucose lowering | 11
  Diuretics | 11
  Analgesics | 9
  Calcium Channel Blockers | 8
  ACE Inhibitors | 5
  Mineral Supplements | 5
  Antidepressants | 4
  Corticosteroids | 4
  Drugs for treatment of bone disease | 4
  HMG COA Reductase Inhibitors | 4
  Anti-anemic | 3
  Antibacterials | 3
  Antithrombotic | 3
  Dermatologicals | 3
  Drugs for Constipation | 3
  Immunosuppressive agents | 3
  Anti-asthmatics | 2
  Insulin and Analogues | 2
  Anti-andrenergic Antihypertensives | 1
  Anti-arrhythmics | 1
  Antidiarrheals | 1
  Anti-inflammatory/antirheumatic products | 1
  Antineoplastic,immunomodulating agents, cytostatic | 1
  Antipsychotics | 1
  Antivirals for HIV, combinations | 1
  Antivirals, reverse transcriptase inhibitors HIV | 1
  Benzodiazepine derivatives | 1
  Bile therapy | 1
  Blood substitutes/perfusion solutions | 1
  Hemostatics/vitamin K | 1
  Lipotropics | 1
  Other antivirals, HIV treatment | 1
  Other Sex hormones | 1
  Vasoprotectives | 1

ADVERSE EVENTS:
Time Frame: Safety was assessed only as treatment emergent adverse events (TEAEs) as recorded by the treating physician. TEAEs were collected after the first dose of study drug through 30 days after last dose of study drug.
Description: TEAEs were defined as any adverse event (AE) with onset date after the first dose of study drug until 30 days after last dose of study drug. Serious adverse events were reported to AbbVie from the time the physician obtained the participant's informed consent form until 30 days or 5 half-lives following the intake of the last dose of physician-prescribed treatment.
Groups:
- ABBVIE REGIMEN: ABBVIE REGIMEN: ombitasvir/paritaprevir/ritonavir with or without dasabuvir for 12 or 24 weeks in Hepatitis C Virus Genotype 1 (HCV + GT1) participants according to standard of care within local label recommendations for their specific disease characteristics (cirrhotic status, genotype).
- ABBVIE REGIMEN Plus Ribavirin (RBV): ABBVIE REGIMEN plus ribavirin (RBV): ombitasvir/paritaprevir/ritonavir with or without dasabuvir and with weight-based RBV for 12 or 24 weeks in HCV + GT1 participants according to standard of care within local label recommendations for their specific disease characteristics (cirrhotic status, genotype).
Arm/Group | ABBVIE REGIMEN | ABBVIE REGIMEN Plus Ribavirin (RBV)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/16
Serious Adverse Events (participants affected / at risk) | 5/49 | 2/16
Other Adverse Events (participants affected / at risk) | 5/49 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBVIE REGIMEN (N=49) | ABBVIE REGIMEN Plus Ribavirin (RBV) (N=16)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC FIBROSIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATOTOXICITY (Hepatobiliary disorders) | 1 (1) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0)
PERITONITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBVIE REGIMEN (N=49) | ABBVIE REGIMEN Plus Ribavirin (RBV) (N=16)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1)
TREATMENT FAILURE (General disorders) | 0 (0) | 1 (1)
HEPATITIS C (Hepatobiliary disorders) | 0 (0) | 1 (1)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT02851069/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT02851069/SAP_001.pdf